# Electrical Activation Mapping Guided Tailor Made Approach for Cardiac Resynchronization Therapy

# 1.0 BACKGROUND

Cardiac resynchronization therapy (CRT) is an established therapy for symptomatic heart failure patients despite optimal medical therapy with prolongation of QRS duration on surface electrocardiogram. Several pivotal studies have demonstrated a significant benefit in terms of mortality and morbidity in patients described above.<sup>1-7</sup> However, there are still 30 to 40% of studied patients being nonresponder to CRT, despite its proven benefit. The responder rate is particular poor in patients with non-LBBB pattern of conduction disturbance<sup>8-15</sup> with one recent study showing non-LBBB patients has a responder rate of only 38%. 15 The plausible reasons of lack of effect of CRT in these patients include relative less baseline electrical dyssynchrony, a homogenous type of conduction delay without a discrete line of block, lack of electrical ventricular uncoupling and inability to improve or even in some case worsening of electrical dyssynchrony with CRT.<sup>15-21</sup>The electrical activation response to conventional CRT varies between individual patients may not be predicted by baseline conduction disturbance. 10,17,19,22 The prevalence of non-LBBB type of conduction disturbance is reported to be as high as 44% in heart failure patients with increase in QRS duration.<sup>23</sup> Hence, a large proportion of heart failure patients with prolonged QRS duration will not benefit from CRT.

The quest to improve CRT responder rate has been subject of intense research interest. Apart from screening for subgroup of heart failure patients with better responder rate to conventional CRT, another possibility is to improve the efficacy of current CRT delivery system. There are two major approaches that have been studied to improve CRT delivery namely selecting the optimal site for LV pacing and alternate method of CRT delivery other than pacing at single epicardial LV site. Study have demonstrated that targeting the LV lead to the site of latest mechanical contraction as determined by strain echocardiogram improved the responder rate.<sup>24</sup> Other studies looks into local electrogram guided placement of LV lead to the latest electrically activated segment inside coronary sinus branch.<sup>25</sup>Regarding alternate way of CRT delivery, there are interests in using direct His-bundle pacing to overcome the longitudinal conduction delay in the His-Purkinjie system. It has been shown that significant narrowing of QRS duration and favorable clinical outcome when compare to conventional CRT can be achieved with direct Hisbundle pacing.<sup>26</sup> Intuitively, direct-His bundle pacing may provide benefit over pre-excitation of the left ventricle by conventional CRT in patients with right bundle branch block (RBBB) pattern of conduction disturbance. Other potential method to improve CRT outcome is the delivery of multipoint pacing (two LV sites together with one RV site and two RV sites together with one LV site) by recruiting more myocardium to contract simultaneously. 27-29 Pacing the LV endocardium as compared to epicardium via a coronary access has been shown to improve acute hemodynamic response but however there is no long-term clinical result of endocardial LV pacing comparing to epicardial LV pacing.<sup>30</sup>

The ability to deliver CRT using different configuration provides opportunity to tailor made resynchronization therapy to heterogenous group of patient in terms of activation delay. This is in contrary to the current concept of a single configuration of CRT deliver suit all patients with widening of QRS duration disregard of pattern of activation delay. Hence the aim of our study is to

investigate whether there is an optimal configuration of CRT delivery that varies between patients with different pattern of activation delay.

Previous study on noninvasive activation pattern has shown that responders showed higher degree of baseline dyssynchrony and greater improvement of dyssynchrony by CRT when compared to nonresponders. The optimal configuration of CRT delivery is defined by that result in the greatest improvement of electrical dyssynchrony. The acute change in electrical dyssynchrony indices will be compare between the optimal configuration and the conventional configuration, namely biventricular pacing with single LV lead in posterior or lateral branch of coronary sinus. A significant different between the two configurations would suggest that there indeed is an optimal configuration of CRT delivery and a tailor made strategy is feasible. To prove this concept of tailor made strategy, devices will be implanted to deliver CRT using the optimal configuration determined by noninvasive electrical activation mapping in non-LBBB patients. The medium term improvement of surrogate marker of LV systolic volume will be compared to that of a predefined level of 40%.

Our group has been using echocardiogram to study mechanical dyssynchrony in patients with heart failure and pacing induced LV dysfunction in predicting response to CRT.31-47 However, in subsequent multi-center trial studying 12 different echocardiographic parameters of mechanical dyssynchrony in predicting CRT response, no single echocardiographic measure of dyssynchrony was shown to improve patient selection for CRT.<sup>48</sup> The results of the study further strengthen the concept that the response to conventional CRT therapy cannot be predicted by baseline dyssynchrony pattern. It is rather the degree of improvement from baseline that will predict response to CRT therapy. The degree of dyssynchrony improvement on the other hand is determined by the interaction of baseline electrical substrate and the activation change brings about by CRT. The electrical substrate is fixed but different configuration of CRT delivery, including different location of LV lead, can produce different changes in activation. In order to study the interaction of electrical substrate and change in activation brings about by CRT, a tool that allows global electrical mapping of both the LV and RV is considered to be important not only to elucidate important information like location of conduction block but also to study the interaction of the left and right ventricle. 17-19,22

# 2.0 STUDY OBJECTIVES

The purpose is to prospectively study the feasibility to optimize configuration of CRT delivery for acute correction of electrical dyssynchrony using a noninvasive mapping of global electrical activation.

#### **Study Hypothesis**

Tailor-made configuration of CRT delivery is feasible and able to improve responder rate compare to single method of CRT delivery in candidates with known poor response to CRT.

## Primary outcome measure

Responder rate of greater than 10% of LV end systolic volume reduction in patients undergoing tailor-made approach of CRT delivery at 6 months. The responder rate is to compare with pre-defined level of 40% for single method of CRT delivery namely biventricular pacing with LV lead in coronary sinus.

## **Secondary outcome measures**

- 1. The acute electrical dyssynchrony indices of different methods of CRT delivery.
- 2. The hemodynamic responses of different methods of CRT delivery.
- 3. Procedure duration and implantation success rate of the optimal CRT delivery method as determined by the best improvement in electrical dyssynchrony indices.
- 4. Cine images (PA, LAO 30°, RAO 30°) and Chest X ray (PA view)
- 5. Peri-operative and 6 months follow-up complications rate:
  - a. Thromboembolic event
  - b. Dislodgement and migration of pacing leads
  - c. Phrenic nerve stimulation
  - d. Others
- 6. Echocardiogram parameters at baseline and 6 months: left ventricular systolic and diastolic volume, left ventricular ejection fraction, degree of mitral regurgitation, strain imaging.
- 7. NYHA class, 6 minute hall walk test and quality of life using Minnesota's questionnaire at baseline and 6 months.
- 8. Electrical parameters including threshold, sensitivity and lead impedance of pacing leads at implant and 6 months follow-up.

#### 3.0 PATIENT SELECTION CRITERIA

#### Inclusion criteria:

Adult (aged 18 or above) of both sexes
Ischemic or non-ischemic cause of heart failure
QRS duration > 120 ms, non -LBBB type of conduction disturbance
NYHA class III or above
Sinus rhythm
Informed consent by the patient

Already received stable dose of guideline directed medical therapy for at least 3 months

#### **Exclusion criteria**

LBBB\* patients

Pregnant women

Participation in another study

Patient with contraindication to left ventricle catheterization by a retrograde aortic approach (eg mechanical aortic valve, severe aortic stenosis and aortic dissection)

\*The definitions of LBBB (QRS duration ≥130 ms; QS or rS in lead V1; broad R waves in leads I, aVL, V5, or V6; and absent q waves in leads I, V5, and V6).

#### 4.0 STUDY DESIGN

This is a prospective, single-center, non-randomized study, aiming to demonstrate the feasibility of tailor-made CRT delivery to optimize electrical dyssynchrony correction using noninvasive study of electrical activation in subgroup of patients with poor response to CRT.

Study will be performed in accordance with Declaration of Helsinki.

#### **Recruitment Method**

Patients with relative narrow QRS complex and non-LBBB pattern of conduction disturbance who is referred for CRT therapy will be recruited for the study. The clinical care of the patients recruited will not be different to other patients receiving CRT. The study will be carried out in Prince of Wales Hospital, Hong Kong.

#### 5.0 STATISTICAL CONSIDERATION

## **Hypothesis**

The null and alternative hypotheses are as follows:

H0: The responder rate of tailor-made approach  $\leq 40\%$ 

HA: The responder rate of tailor-made approach > 40%

Sample size was calculated employing binomial methods with the following assumptions were used:

Expected responder rate for tailor-made approach =60% Historical control responder rate =40% Test significance level (a) = 0.05 (1-sided) Power= 80%

Based on the above assumptions, the sample size was calculated as 77. Accounting for the attrition of 20%, the total required sample size is 93 patients with device implanted.

# Statistical method for additional analysis

All continuous data will be summarized with the number of non-missing data, mean ± standard deviation, median and range (minimum – maximum). T test will be used for the comparison between the groups. In case the assumption for t test is violated, then the equivalent nonparametric test, such as Wilcoxon rank sum test, Kolmogorov-smirnov test, will be used instead. The normality assumption will be tested by the normality test with the aid of QQ plot.

All categorical data will be tabulated with number of occurrence and percentage. Chi-square test will be used for the comparison between the groups. In case the expected counts in each cell is less than 5, then Fisher's exact test will be used instead.

## Procedures for reporting any deviation(s) from the original statistical plan

Any deviations from the statistical analysis plan will be documented.

The treatment of missing, unused or spurious data, including drop-outs and withdrawals.

No imputation techniques will be used.

# 6.0 PROTOCOL DESCRIPTION

#### Patient informed consent

The investigator is responsible for obtaining informed consent from each prospective study patient prior to the performance of any study related procedures. After a patient has been provided with the information of the study and given time to think on whether to participating into the study, the patient will be asked to sign and date a consent form. One copy of the signed patient consent form must be handed out to the patient and one must be filed by the investigator in the investigator files. After the patient and the investigator have signed and dated the consent form, the study data collection process may start.

Patients meeting all the inclusion criteria and not meeting any of the exclusion criteria are eligible for the study. Data will be collected at the following study visits:

Enrollment

Noninvasive electrical activation and acute hemodynamic study

Pre-discharge (PDH) (≤ 72 hours post implant)

Month 3 follow-up visit: 90 ± 14 days post implant Month 6 follow-up visit: 180 ± 14 days post implant

Table 1. Data collection for each scheduled visit

| | Enrollment | Implant | PDH* | Month | Month |
|----------------------|------------|---------|------|-------|-------|
| | | * | | 3 | 6 |
| Patient Informed | X | | | | |
| Consent | | | | | |
| Echocardiogram | X | | X | X | X |
| Medical History | X | | | | |
| Cardiovascular | X | X | X | X | X |
| Medication | | | | | |
| NYHA Class | X | | | X | X |
| 6MHW | X | | | X | X |
| SF-36QoL | X | | | X | X |
| 12-lead | X | X | | X | X |
| electrocardiogram | | | | | |
| Cine images | | X | | | |
| Device Interrogation | · | X | X | X | X |
| Adverse Event | X | X | X | X | X |
| Protocol Deviation | X | X | X | X | X |

Figure 1. Study Flow Chart



## Noninvasive mapping of electrical activation

Ventricular activation maps will be acquired simultaneously with hemodynamic measurements using noninvasive mapping system (ECVUE, Medtronic Inc, USA). A thoracic computed tomographic scan will be acquired with the electrodes attached to the patient. Local ventricular activation times will be defined as the onset of the QRS complex or the pacing spike to the maximal negative slope of each unipolar electrogram.

The following electrical dyssynchrony indices will be derived

- i) Total activation time (TAT) is defined as the time difference between the earliest and latest site of activation on the entire ventricular epicardium (LV and RV);
- ii) RVTAT is defined as the time difference between the earliest and latest site of activation on the RV ventricular epicardium;
- iii) LVTAT is defined as the time difference between the earliest and latest site of activation on the LV ventricular epicardium;
- iv) Ventricular electrical uncoupling (VEU) is defined as mean LV activation time minus mean RV activation time (LVTAT-RVTAT)
- v) Intra-LV electrical dyssynchrony index (ED) is the standard deviation of activation times at 500 sites on the LV epicardium, including the epicardial aspect of the septum.

## Placement of electrophysiology catheters for CRT delivery

Pacing leads will be placed in high right atrium, His-bundle region, right ventricular apex, high septal RV, coronary sinus posterior/lateral branch, coronary sinus anterior branch, lateral and septal region of endocardial LV in order to deliver CRT in 8 different configurations as stated below:

- 1) Conventional biventricular pacing with RV lead in right ventricular apex and LV lead in lateral or posterior branch of coronary sinus
- 2) Biventricular pacing with the LV lead in coronary sinus in closest possible proximity to the latest electrical activation region (18 region) if it is different to the site tested in (1)
- 3) Direct His-bundle pacing
  - i) His bundle pacing catheter distal tip as cathode and RV lead proximal pole as anode
  - ii) His bundle pacing catheter distal tip as cathode and proximal pole of LV lead placed in lateral or posterior branch of coronary sinus as anode.
  - iii) His bundle pacing catheter distal tip as cathode and His bundle pacing catheter proximal pole as anode.

## In subjects in sinus rhythm

i) together with RV bipolar pacing with RV lead in RV apex.

# In subjects in AF

i) together with RV bipolar and LV bipolar pacing

## 4) Multi-point pacing

- i) Triple site pacing with two RV leads in the RV apex and high RV septum and LV lead in posterior or lateral branch of coronary sinus.
- ii) Triple site pacing with RV lead in the RV apex and one LV lead in posterior or lateral branch of coronary sinus and the other LV lead in anterior branch of coronary sinus.
- iii) Triple site pacing with RV lead in RV apex and one quadripolar LV lead in posterior or lateral branch of coronary sinus and pacing at 2 sties stimultaneously from the quadripolar lead.

During delivery of CRT the output will be set at twice the capture threshold and pacing impulse will be deliver in VDD mode with an AV delay of 80msec and VV delay at 0msec for all leads in the ventricles.

## Acute hemodynamics studies

Invasive LV hemodynamic measurements of LV dP/dt will be recorded using a micromanometer (Radi Medical Systems, St Jude Medical, USA) placed in the LV cavity.

All measurements will be made with an average of 10 second recordings with no occurrence of premature atrial or ventricular beats during the recording and 1 minute interval between changes in pacing settings.

During sinus rhythm and the 7 configurations of CRT pacing as stated above both noninvasive electrical activation map and acute hemodynamic measurement will be recorded for analysis.

#### **Implantation of CRT device**

1) Conventional pacing configuration

The CRT system will be implanted with standard technique for conventional pacing configuration. Only market released CRT devices and leads will be implanted.

2) Epicardial LV pacing in the latest activation site

LV lead will be placed in the LV latest activation site or the site in closest proximity to the latest activation site and if necessary quadripolar or active fixation LV lead will be used to achieve stability.

# 3) Direct His-bundle pacing

# i) In subjects in sinus rhythm

For direct-His bundle pacing, standard techniques will be use to place an LV lead preferably in the posterolateral branch of the coronary sinus system, RV and right atrial lead. His pacing lead (SelectSecure, model 3830, Medtronic Inc, USA) supported using a dedicated delivery sheath (model C315, Medtronic Inc, USA) or a deflectable lead delivery sheath (model C304, Medtronic Inc, USA) to the site showing His bundle signal on the mapping catheter. Multiple position to optimize QRS narrowing and threshold could be tested. The His pacing lead and the LV lead will be connected via a Y-adapter (model 5866-38M, Medtronic Inc, USA). The HBP will be connected to the cathode and the LV tip to the anode of the Y-connector.

#### ii) In subjects in AF

The same as for subjects in sinus rhythm except the His pacing lead will be connected to the atrial port of the CRT device and LV lead into the LV port of the CRT device without the use of a Y adapter.

## 4) Multiple point pacing

For multiple point pacing, the septal RV and the bipolar LV leads will be connected to the LV port using a parallel Y-adapter (model 2872, Medtronic Inc, USA) for the 2 RV leads group. Whilst the anterior bipolar and posterior/lateral LV lead will be connected using a parallel Y-adapter (model 2872, Medtronic Inc, USA) for the 2 LV leads group. If simultaneous pacing from 2 sites o fthe quadripolar LV lead pacing is the optimal configuration, a quadripolar lead will be connected to the LV port.

# **CRT** programming

| Para meter | Mandatory Device Setting |
|---|---|
| Mode | DDD or DDDR |
| Base Rate | ≤ 60 min-1 |
| Max. Sensor Rate/Max.<br>Tracking Rate | 140 min-1 |
| Mode Switch | "On" if atrial tachyarrhythmia are suspected |
| Paced AV Delay | 150 ms |

| Sensed AV Delay | 120 ms |
|-----------------|--------|
| V-V Delay | 0ms |

#### **Adverse Events**

#### **Definition**

**Adverse Event (AE)** is defined as any untoward medical occurrence in a patient who participates in a clinical investigation. This definition does not imply that there is a relationship between adverse event and the clinical investigation.

# **Serious Adverse Event (SAE)** is defined as an adverse event that

- a) led to death
- b) led to a serious deterioration in the health of the subject that
- i. resulted in a life-threatening illness or injury
- ii. resulted in a permanent impairment of a body structure or a body function
- iii. requiredin-patienthospitalizationorprolongationofexistinghospitalization
- iv. resulted in medical or surgical intervention to prevent permanent impairment to
- c) led to body structure or a body function to foetal distress, foetal death or a congenital abnormality or birth defect .

# **List of Anticipated Adverse Events**

Possible adverse events (in alphabetical order) associated with the acute noninvasive activation mapping and hemodynamic study, include, but are not limited to the following:

- Air embolism
- Allergic reaction
- Arterial or venous occlusion
- Arterial, venous or cardiac perforation
- Asystole
- Bleeding
- Cardiac tamponade
- Death
- Erosion
- Exacerbation of heart failure
- Infection

- Myocardial damage
- Thromboembolism

Possible adverse events (in alphabetical order) associated with the CRT device implantation, include, but are not limited to the following:

Acceleration of arrhythmias (caused by device)

Angina pectoris

Air embolism

Allergic reaction

Asystole

Bleeding

Cardiac tamponade

Chronic nerve damage

Death

Erosion

Exacerbation of heart failure

Excessive fibrotic tissue growth

Extracardiac stimulation (phrenic nerve, diaphragm, chest wall)

Extrusion

Fluid accumulation

Formation of hematomas or cysts

Histotoxic reaction

Infection

Loss of capture

Myocardial damage

Oversensing / undersensing

Palpitations due to documented arrhythmias

Phrenic nerve stimulation

Pneumothorax

Thromboembolism

Venous occlusion

Venous or cardiac perforation

# **Adverse Events Recording and Reporting**

Safety surveillance and reporting will be done for all patients enrolled in the study. This will be started from the time patient provides with the informed consent until the last study visit has been performed or the patient has died or the patient concludes his participation into the study.

All **Serious Adverse Event** is to be documented and reported to the research ethics committee within 24 hours of notification.

As soon as the final details are available for the AE, the information should be reported on the AE case report form:

- Hospitalization details (if applicable)
- Diagnostic test information (if applicable)
- Treatment given (if applicable)
- Final medical diagnosis and cause
- Patient condition
- Final AE status
- Seriousness of AE based on final medical diagnosis and cause
- Relationship of AE to clinical investigation based on final medical diagnosis and cause

# **Study Termination**

All reasonable efforts should be made to retain the patient in the clinical investigation until completion of the clinical investigation.

If a patient concludes their participation in the study, the future care and management will not be affected, whether it is voluntary or otherwise:

- A patient completes the study (Month 6 follow-up).
- A patient / family member may request to withdraw from the clinical investigation at any time with no effect to the patient's present care.
- A patient dies.
- An investigator may withdraw a patient from the study at any time as according to the best interest to the patient.

## Risks associated with Participation in the Clinical Investigation

The risks involved with this study are comparable to those associated with the implant of any CRT.

The additional risks are related to the computerized tomography of the heart with possible complication of contrast injury to kidney and allergic reaction. Other additional risks are related to pre-implantation electrical activation study which involves putting in pacing catheters and pressure monitoring catheters in the body with possible risk of injury to the heart, blood vessel, bleeding, wound complications and infection.

#### **Risk Minimization Actions**

Additional risks may exist. Risks can be minimized through compliance with this CIP, performing procedures in the appropriate hospital environment, adherence to subject selection criteria, close monitoring of the subject's physiologic status during research procedures and/or follow-ups.

## **Anticipated Benefits**

The proposed tailor made method of CRT delivery may improve the outcome inpatient that will be recruited in the study with high incident of non responding to CRT by improving electrical dyssynchrony correction.

#### REFERECES

- 1. Bristow, M.R., Saxon, L.A., Boehmer, J. et al, Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004;350:2140–2150.
- 2. Cleland, J.G., Daubert, J.C., Erdmann, E. et al, The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005;352:1539–1549.
- 3. Tang, A.S.L., Wells, G., Talajic, M. et al, Cardiac-resynchronization therapy for mild-to-moderate heart failure. N Engl J Med. 2010;363:2385–2395.
- 4. Bradley, D.J., Bradley, E.A., Baughman, K.L. et al, Cardiac resynchronization and death from progressive heart failure: a meta-analysis of randomized controlled trials. JAMA. 2003;289:730–740.
- 5. Cleland JG, Abraham WT, Linde C, Gold MR, Young JB, Claude Daubert J, Sherfesee L, Wells GA, Tang AS. An individual patient meta-analysis of five randomized trials assessing the effects of cardiac resynchronization therapy on morbidity and mortality in patients with symptomatic heart failure. Eur Heart J 2013;34:3547–3556.
- 6. Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, et al. ESC guidelines on cardiac pacing and cardiac resynchronization therapy: the task force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA). Europace 2013;15(8):1070–118.
- 7. Russo AM, Stainback RF, Bailey SR, Epstein AE, Heidenreich PA, Jessup M, et al. ACCF/HRS/AHA/ASE/HFSA/SCAI/SCCT/SCMR 2013 appropriate use criteria for implantable cardioverter–defibrilla- tors and cardiac resynchronization therapy: a report of the American College of Cardiology Foundation appropriate use criteria task force, Heart Rhythm Society, American Heart Association, American Society of Echocardiography, Heart Failure Society of America, Society for Cardiovascular Angiography and Interventions, Society of Cardiovas- cular Computed Tomography, and Society for Cardiovascular Magnetic Resonance. J Am Coll Cardiol 2013;61(12):1318–68.

- 8. Sipahi, I., Chou, J.C., Hyden, M., Rowland, D.Y., Simon, D.I., Fang, J.C. Effect of QRS morphology on clinical event reduction with cardiac resynchronization therapy: meta-analysis of randomized controlled trials. Am Heart J. 2012;163:260–267
- 9. Peterson, P.N., Greiner, M.A., Qualls, L.G. et al, QRS duration, bundle-branch block morphology, and outcomes among older patients with heart failure receiving cardiac resynchronization therapy. JAMA. 2013;310:617–626.
- 10. Eschalier R, Ploux S, Ritter P, Haïssaguerre M, Ellenbogen KA, Bordachar P.Nonspecific intraventricular conduction delay: Definitions, prognosis, and implications for cardiac resynchronization therapy. Heart Rhythm. 2015 May;12(5):1071-9.
- 11. Nery PB, Ha AC, Keren A, Birnie DH. Cardiac resynchronization therapy in patients with left ventricular systolic dysfunction and right bundle branch block: a systematic review. Heart Rhythm 2011;8 (7):1083–7.
- 12. ByrneMJ,HelmRH,DayaS,OsmanNF,HalperinHR,BergerRD,etal. Diminished left ventricular dyssynchrony and impact of resynchronization in failing hearts with right versus left bundle branch block. J Am Coll Cardiol 2007;50(15):1484–90.
- 13. Zareba, W., Klein, H., Cygankiewicz, I. et al, CRT effectiveness by QRS duration and morphology in the MADIT-CRT patients. Heart Rhythm. 2010;7:24–25.
- 14. Gold MR, Thébault C, Linde C, Abraham WT, Gerritse B, Ghio S, St John Sutton M, Daubert JC. Effect of QRS duration and morphology on cardiac resynchronization therapy outcomes in mild heart failure: results from the Resynchronization Reverses Remodeling in Systolic Left Ventricular Dysfunction (REVERSE) study. Circulation. 2012 Aug 14;126(7):822-9.
- 15. Hara H, Oyenuga OA, Tanaka H, Adelstein EC, Onishi T, McNamara DM, Schwartzman D, Saba S, Gorcsan J 3rd. The relationship of QRS morphology and mechanical dyssynchrony to long-term outcome following cardiac resynchronization therapy. Eur Heart J. 2012 Nov;33(21):2680-91.
- 16. Haghjoo, M., Bagherzadeh, A., Farahani, M., Haghighi, Z.O., Sadr-Ameli, M.A. Significance of QRS morphology in determining the prevalence of mechanical dyssynchrony in heart failure patients eligible for cardiac resynchronization: particular focus on patients with right bundle branch block with and without coexistent left-sided conduction defects. Europace. 2008;10:566–571.
- 17. Ghosh S, Silva JN, Canham RM, Bowman TM, Zhang J, Rhee EK, Woodard PK, Rudy Y. Electrophysiologic substrate and intraventricular left ventricular

- dyssynchrony in nonischemic heart failure patients undergoing cardiac resynchronization therapy. Heart Rhythm. 2011 May;8(5):692-9.
- 18. Ploux S, Eschalier R, Whinnett ZI, Lumens J, Derval N, Sacher F, Hocini M, Jaïs P, Dubois R, Ritter P, Haïssaguerre M, Wilkoff BL, Francis DP, Bordachar P. Electrical dyssynchrony induced by biventricular pacing: implications for patient selection and therapy improvement. Heart Rhythm. 2015 Apr;12(4):782-91
- 19. Ploux, S., Lumens, J., Whinnett, Z. et al, Noninvasive electrocardiographic mapping to improve patient selection for cardiac resynchronization therapy: beyond QRS duration and left bundle branch block morphology. J Am Coll Cardiol. 2013;61:2435–2443.
- 20. Auricchio, A., Fantoni, C., Regoli, F., Carbucicchio, C., Goette, A., Geller, C., Kloss, M., Klein, H. Characterization of left ventricular activation in patients with heart failure and left bundle-branch block. Circulation. 2004;109:1133–1139.
- 21. Auricchio A, Lumens J, Prinzen FW. Does cardiac resynchronization therapy benefit patients with right bundle branch block: cardiac resynchronization therapy has a role in patients with right bundle branch block. Circ Arrhythm Electrophysiol. 2014 Jun;7(3):532-42.
- 22. Varma N, Jia P, Rudy Y. Electrocardiographic imaging of patients with heart failure with left bundle branch block and response to cardiac resynchronization therapy. J Electrocardiol. 2007 Nov-Dec;40(6 Suppl):S174-8.
- 23. Lund LH, Jurga J, Edner M, Benson L, Dahlström U, Linde C et al Prevalence, correlates, and prognostic significance of QRS prolongation in heart failure with reduced and preserved ejection fraction. Eur Heart J 2013;34:529–539
- 24. Khan FZ, Virdee MS, Palmer CR, Pugh PJ, O'Halloran D, Elsik M, Read PA, Begley D, Fynn SP, Dutka DP. Targeted left ventricular lead placement to guide cardiac resynchronization therapy: the TARGET study: a randomized, controlled trial. J Am Coll Cardiol. 2012 Apr 24;59(17):1509-18.
- 25. Gold MR, Birgersdotter-Green U, Singh JP, Ellenbogen KA, Yu Y, Meyer TE, Seth M, Tchou PJ. The relationship between ventricular electrical delay and left ventricular remodelling with cardiac resynchronization therapy. Eur Heart J. 2011 Oct;32(20):2516-24
- 26. Lustgarten DL, Crespo EM, Arkhipova-Jenkins I, Lobel R, Winget J, Koehler J, Liberman E, Sheldon T. His-bundle pacing versus biventricular pacing in cardiac resynchronization therapy patients: A crossover design comparison. Heart Rhythm. 2015 Jul;12(7):1548-57.

- 27. Anselme F, Bordachar P, Pasquié JL, Klug D, Leclercq C, Milhem A, Alonso C, Deharo JC, Gras D, Probst V, Piot O, Savouré A. Safety, feasibility, and outcome results of cardiac resynchronization with triple-site ventricular stimulation compared to conventional cardiac resynchronization. Heart Rhythm. 2016 Jan;13(1):183-9
- 28. Lenarczyk R, Kowalski O, Sredniawa B, Pruszkowska-Skrzep P, Mazurek M, Jędrzejczyk-Patej E, Woźniak A, Pluta S, Głowacki J, Kalarus Z. Implantation feasibility, procedure-related adverse events and lead performance during 1-year follow-up in patients undergoing triple-site cardiac resynchronization therapy: a substudy of TRUST CRT randomized trial. J Cardiovasc Electrophysiol. 2012 Nov;23(11):1228-36.
- 29. Bordachar P, Alonso C, Anselme F, Boveda S, Defaye P, Garrigue S, Gras D, Klug D, Piot O, Sadoul N, Leclercq C. Addition of a second LV pacing site in CRT nonresponders rationale and design of the multicenter randomized V(3) trial. J Card Fail. 2010 Sep;16(9):709-13.
- 30. Morgan JM, Biffi M, Gellér L, Leclercq C, Ruffa F, Tung S, Defaye P, Yang Z, Gerritse B, van Ginneken M, Yee R, Jais P; ALSYNC Investigators. Atternate Site Cardiac ResynChronization (ALSYNC): a prospective and multicentre study of left ventricular endocardial pacing for cardiac resynchronization therapy. Eur Heart J. 2016 Jan 18. pii: ehv723.
- 31. Fang F, Zhang Q, Chan JY, Razali O, Azlan H, Chan HC, Sanderson JE, Xie JM, Yu CM. Early pacing-induced systolic dyssynchrony is a strong predictor of left ventricular adverse remodeling: Analysis from the Pacing to Avoid Cardiac Enlargement (PACE) trial. Int J Cardiol. 2012.
- 32. Zhang Q, van Bommel RJ, Chan JYS, Delgado V, Liang Y, Schalij MJ, Bax JJ, Fang F, Yip GW, Yu CM. Diverse patterns of longitudinal and radial dyssynchrony in patients with advanced systolic heart failure. Heart 2011 Apr;97(7):574-8.
- 33. Fang F, Chan JYS, Yip GW, Xie JM, Zhang Q, Fung JW, Lam YY, Yu CM. Prevalence and determinants of left ventricular systolic dyssynchrony in patients with normal ejection fraction received right ventricular apical pacing: a real-time three-dimensional echocardiographic study. Eur J Echocardiogr. 2010 Mar;11(2):109-18.
- 34. Zhang Q, van Bommel RJ, Fung JW, Chan JYS, Bleeker GB, Ypenburg C, Yip G, Liang YJ, Schalij MJ, Bax JJ, Yu CM. Tissue Doppler velocity is superior to strain imaging in predicting long-term cardiovascular events after cardiac resynchronisation therapy. Heart. 2009 Jul;95(13):1085-90.

- 35. Zhang Q, Fang F, Yip GW, Chan JYS, Shang Q, Fung JW, Chan AK, Liang YJ, Yu CM. Difference in prevalence and pattern of mechanical dyssynchrony in left bundle branch block occurring in right ventricular apical pacing versus systolic heart failure. Am Heart J. 2008 Nov;156(5):989-95.
- 36. Fung JW, Lam YY, Zhang Q, Yip GW, Chan WW, Chan GC, Chan JYS, Yu CM. Effect of left ventricular lead concordance to the delayed contraction segment on echocardiographic and clinical outcomes after cardiac resynchronization therapy. J Cardiovasc Electrophysiol. 2009 May;20(5):530-5.
- 37. Zhang Y, Yip GW, Chan AK, Wang M, Lam WW, Fung JW, Chan JYS, Sanderson JE, Yu CM. Left ventricular systolic dyssynchrony is a predictor of cardiac remodeling after myocardial infarction. Am Heart J. 2008 Dec;156(6):1124-32.
- 38. Zhang Q, Fung JW, Chan JYS, Yip G, Lam YY, Liang YJ, Yu CM. Difference in long-term clinical outcome after cardiac resynchronisation therapy between ischaemic and non-ischaemic aetiologies of heart failure. Heart. 2009 Feb;95(2):113-8.
- 39. Zhang Q, Fung JW, Yip GW, Chan JYS, Lee AP, Lam YY, Wu LW, Wu EB, Yu CM. Improvement of Left Ventricular Myocardial Short-axis, but not Longaxis Function or Torsion after Cardiac Resynchronization Therapy-An Assessment by Two-Dimensional Speckle Tracking. Heart. 2008 Jan 15.
- 40. Van de Veire NR, Yu CM, Ajmone-Marsan N, Bleeker GB, Ypenburg C, De Sutter J, Zhang Q, Fung JW, Chan JYS, Holman ER, van der Wall EE, Schalij MJ, Bax JJ. Triplane tissue Doppler imaging: a novel three-dimensional imaging modality that predicts reverse left ventricular remodelling after cardiac resynchronisation therapy. Heart. 2008 Mar;94(3):e9.
- 41. Yu CM, Gorcsan J 3rd, Bleeker GB, Zhang Q, Schalij MJ, Suffoletto MS, Fung JW, Schwartzman D, Chan JYS, Tanabe M, Bax JJ. Usefulness of tissue Doppler velocity and strain dyssynchrony for predicting left ventricular reverse remodeling response after cardiac resynchronization therapy. Am J Cardiol. 2007 Oct 15;100(8):1263-70.
- 42. Fung JW, Chan JYS, Yip GW, Chan HC, Chan WW, Zhang Q, Yu CM. Effect of left ventricular endocardial activation pattern on echocardiographic and clinical response to cardiac resynchronization therapy. Heart. 2007 Apr;93(4):432-7.
- 43. Yu CM, Chan JYS, Zhang Q, Yip GW, Chan CK, Kum LC, Wu L, Lee AP, Lam YY, Fung JW. Benefits of cardiac resynchronization therapy for heart failure patients with narrow QRS complexes and coexisting systolic asynchrony by echocardiography. J Am Coll Cardiol. 2006 Dec 5;48(11):2251-7.

- 44. Yu CM, Zhang Q, Yip GW, Chan JYS, Lee PW, Wu LW, Lam YY, Kum LC, Chan HC, Chan S, Fung JW. Are left ventricular diastolic function and diastolic asynchrony important determinants of response to cardiac resynchronization therapy? Am J Cardiol. 2006 Oct 15;98(8):1083-7.
- 45. Fung JW, Zhang Q, Yip GW, Chan JYS, Chan HC, Yu CM. Effect of Cardiac Resynchronization Therapy in Patients with Moderate Left Ventricular Systolic Dysfunction and Wide QRS Complex: A Prospective Study. J Cardiovasc Electrophysiol. 2006 Sep 20.
- 46. Yu CM, Zhang Q, Fung JW, Chan HC, Chan JYS, Yip GW, Kong SL, Lin H, Zhang Y, Sanderson JE. A novel tool to assess systolic asynchrony and identify responders of cardiac resynchronization therapy by tissue synchronization imaging. J Am Coll Cardiol. 2005 Mar 1;45(5):677-84.
- 47. Zhang Q, Yu CM, Fung JW, Zhang Y, Chan JYS, Chan HC, Yip GW, Sanderson JE. Assessment of the effect of cardiac resynchronization therapy on intraventricular mechanical synchronicity by regional volumetric changes. Am J Cardiol. 2005 Jan 1;95(1):126-9.
- 48. Chung ES, Leon AR, Tavazzi L, Sun JP, Nihoyannopoulos P, Merlino J, Abraham WT, Ghio S, Leclercq C, Bax JJ, Yu CM, Gorcsan J 3rd, St John Sutton M, De Sutter J, Murillo J. Results of the Predictors of Response to CRT (PROSPECT) trial. Circulation. 2008 May 20;117(20):2608-16.